CLINICAL TRIAL: NCT02476760
Title: The Use of Incretin-based Drugs and the Risk of Acute Pancreatitis in Patients With Type 2 Diabetes
Brief Title: Incretin-based Drugs and Acute Pancreatitis
Status: Completed | Type: Observational
Sponsor: Canadian Network for Observational Drug Effect Studies, CNODES (Other)
Collaborators: Drug Safety and Effectiveness Network, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: Q13-06B
Record Dates: First submitted 2015-06-17; First posted 2015-06-19 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Incretins; Antidiabetic agents; Pancreatitis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Pancreatitis | interventions — Dipeptidyl-Peptidase IV Inhibitors; Sitagliptin Phosphate; Vildagliptin; saxagliptin; Glucagon-Like Peptide-1 Receptor Agonists; Exenatide; Liraglutide; Insulins; Injections; Inhalation; Biguanides; Hypoglycemic Agents; Phenformin; Metformin; Buformin; Sulfonylurea Compounds; Glyburide; Chlorpropamide; Tolbutamide; glibornuride; Tolazamide; Carbutamide; Glipizide; gliquidone; Gliclazide; metahexamide; glisoxepide; glimepiride; Acetohexamide; glymidine; Thiazolidinediones; Troglitazone; Rosiglitazone; Pioglitazone; Glycoside Hydrolase Inhibitors; Acarbose; miglitol; voglibose; meglitinide; repaglinide; Nateglinide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Treated with incretins: Current use of incretin-based drugs ((DPP-4 inhibitors [sitagliptin, vildagliptin, and saxagliptin] or GLP-1 analogs [exenatide, liraglutide]) alone or in combination with other anti-diabetic drugs (if the prescription overlaps with the index or event day with a 30-day grace period).
  Interventions: Drug: DPP-4 inhibitors; Drug: GLP-1 analogs
- Treated with insulin: Any use of insulins between base cohort entry and the index or event day (alone or in combination with other antidiabetic drugs) and no current use of incretin-based drugs.
  Interventions: Drug: Insulins
- Treated with ≥2 oral hypoglycemic agents: Current use of 2 or more non-insulin anti-diabetic medications (biguanides, sulfonylureas, thiazolidinediones, alphaglucosidase inhibitors, meglitinides) (if the prescriptions overlap with the index or event day with a 30-day grace period), and no current use of incretin-based drugs or insulins.
  Interventions: Drug: Biguanides; Drug: Sulfonylureas; Drug: Thiazolidinediones; Drug: Alpha-glucosidase inhibitors; Drug: Meglitinides
- Treated with a single oral agent: Current use of any single non-insulin anti-diabetic medication (biguanides, sulfonylureas, thiazolidinediones, alpha-glucosidase inhibitors, meglitinides) (if the prescription overlaps with the index or event day with a 30-day grace period) and no current use of more than 2 OHAs, incretin-based drugs, or insulins from base cohort entry.
  Interventions: Drug: Biguanides; Drug: Sulfonylureas; Drug: Thiazolidinediones; Drug: Alpha-glucosidase inhibitors; Drug: Meglitinides
- Not currently exposed group: All patients not currently exposed to: incretin-based drugs, ≥2 OHAs, a single OHA and no use of insulins since base cohort entry.

INTERVENTIONS:
Drug: DPP-4 inhibitors — Current exposure to DPP-4 inhibitors (ATC A10BH, A10BD07-A10BD13) will be defined as a prescription duration plus a 30-day grace period (to account for non-adherence and the biological half-lives of these drugs) that overlaps with the index day.
  Other Names: incretin-based drugs; sitagliptin; vildagliptin; saxagliptin
  Groups: Treated with incretins
Drug: GLP-1 analogs — Current exposure to GLP-1 analogs (ATC A10BX04, A10BX07) will be defined as a prescription duration plus a 30-day grace
  Other Names: incretin-based drugs; exenatide; liraglutide
  Groups: Treated with incretins
Drug: Insulins — Current exposure to insulin (ATC A10A) will be defined as any use of insulin between base cohort entry and the index day.
  Other Names: insulins and analogues for injection, fast-acting; insulins and analogues for injection, intermediate-acting; insulins and analogues for injection, long-acting; insulins and analogues for inhalation
  Groups: Treated with insulin
Drug: Biguanides — Current exposure to biguanides (ATC A10BA) will be defined as a prescription duration plus a 30-day grace period (to account for non-adherence and the biological half-lives of these drugs) that overlaps with the index day.
  Other Names: oral hypoglycemic agent; phenformin; metformin; buformin
  Groups: Treated with a single oral agent; Treated with ≥2 oral hypoglycemic agents
Drug: Sulfonylureas — Current exposure to sulfonylureas (ATC A10BB or A10BC) will be defined as a prescription duration plus a 30-day grace period (to account for non-adherence and the biological half-lives of these drugs) that overlaps with the index day.
  Other Names: oral hypoglycemic agent; glibenclamide; chlorpropamide; tolbutamide; glibornuride; tolazamide; carbutamide; glipizide; gliquidone; gliclazide; metahexamide; glisoxepide; glimepiride; acetohexamide; glymidine
  Groups: Treated with a single oral agent; Treated with ≥2 oral hypoglycemic agents
Drug: Thiazolidinediones — Current exposure to thiazolidinediones (ATC A10BG) will be defined as a prescription duration plus a 30-day grace period (to account for non-adherence and the biological half-lives of these drugs) that overlaps with the index day.
  Other Names: oral hypoglycemic agent; troglitazone; rosiglitazone; pioglitazone
  Groups: Treated with a single oral agent; Treated with ≥2 oral hypoglycemic agents
Drug: Alpha-glucosidase inhibitors — Current exposure to alpha-glucosidase inhibitors (ATC A10BF) will be defined as a prescription duration plus a 30-day grace period (to account for non-adherence and the biological half-lives of these drugs) that overlaps with the index day.
  Other Names: oral hypoglycemic agent; acarbose; miglitol; voglibose
  Groups: Treated with a single oral agent; Treated with ≥2 oral hypoglycemic agents
Drug: Meglitinides — Current exposure to meglitinides (ATC A10BX02, A10BX03) will be defined as a prescription duration plus a 30-day grace period (to account for non-adherence and the biological half-lives of these drugs) that overlaps with the index (event) day.
  Other Names: oral hypoglycemic agent; repaglinide; nateglinide
  Groups: Treated with a single oral agent; Treated with ≥2 oral hypoglycemic agents

SUMMARY:
The purpose of this study is to determine whether incretin-based drugs (used to treat type 2 diabetes) taken either alone or in combination with other anti-diabetic drugs are associated with an increased risk of acute pancreatitis (AP) compared to other combinations of oral hypoglycemic agents (OHA).

The investigators will carry out separate population based cohort studies using administrative health databases in six jurisdictions in Canada, the US, and the UK. Cohorts will be defined by the initiation of a new anti-diabetic drug when incretin-based drugs entered the market, with follow-up until hospitalization for AP. The results from the separate sites will be combined to provide an overall assessment of the risk of AP in users of incretin-based drugs and by class of incretin-based drugs.

DETAILED DESCRIPTION:
The study objective is to determine whether the use of incretin-based drugs, compared with the use of oral anti-diabetic drug combinations, is associated with an increased risk of acute pancreatitis (AP) in routine clinical practice. A common-protocol approach will be used to conduct retrospective cohort studies using administrative health care data from six jurisdictions (the Canadian provinces of Alberta, Manitoba, Ontario, and Saskatchewan, as well as United States (US) MarketScan and the United Kingdom (UK) Clinical Practice Research Datalink [CPRD]). Briefly, the Canadian databases include population-level data on physician billing, diagnoses and procedures from hospital discharge abstracts, and dispensations for prescription drugs. Ontario data will be restricted to patients aged 65 years and older as prescription data are not available for younger patients. The CPRD is a clinical database that is representative of the UK population and contains the records for patients seen at over 680 general practitioner practices in the UK; these data will be linked to the Hospital Episode Statistics (HES) database, which contains in-hospital diagnosis and procedure data. US MarketScan includes individuals and their dependents covered by large U.S. employer health insurance plans, and government and public organizations.

Study population

In each jurisdiction, the investigators will assemble a base cohort that includes all patients with a first-ever prescription for a non-insulin anti-diabetic drug, including biguanides, sulfonylureas, thiazolidinediones, DPP-4 inhibitors, GLP-1 analogs, alpha-glucosidase inhibitors, meglitinides or combinations of these drugs from the earliest availability of data at each site to the last date of availability of data. The date of prescription (for the CPRD) or dispensation (for all other sites) of the first-ever non-insulin anti-diabetic drug will define the date of base cohort entry. From this base cohort, a study cohort will be created including all patients who initiated a new anti-diabetic drug class during the year in which incretin-based drugs entered the market in each jurisdiction or any time thereafter. These new users consist of both those who are newly-treated for diabetes, as well as those who switch to or add on a new anti-diabetic drug class not included as part of their previous treatment history. The date of study cohort entry is defined by the prescription date of the newly-prescribed drug class. Patients in the study cohort will be followed from the date of study cohort entry until an event (defined below) or censoring due to death, departure from the database, loss of continuous health plan or drug plan enrolment, entry into a long-term care facility, an incident diagnosis of HIV or new prescription of HAART, or the end of the study period (June 30, 2014 or the last date of data availability at that site), whichever occurs first.

Case-control selection

The cohort defined above will be analyzed using a nested case-control analysis, where cases are defined as a hospitalization for AP. Risk set sampling will be used to randomly select up to 20 controls for each case, matched on sex, age (± 365 days), date of study cohort entry (± 180 days), duration of treated diabetes (± 90 days), and duration of follow-up in days.

Exposure assessment

Current exposure to an anti-diabetic drug will be defined as any prescription whose duration plus a 30-day grace period overlaps the index or event date. Current exposure will be classified hierarchically based on the following five mutually-exclusive categories: 1) incretin-based drugs; 2) insulin; 3) ≥2 oral anti-diabetic drugs used in combination therapy; 4) oral anti-diabetic drug monotherapy; and 5) no current exposure to an anti-diabetic drug. Oral anti-diabetic drugs used in combination will serve as the primary reference category as incretin-based drugs are second- to third-line therapy and thus used at a comparable point in the disease management.

Statistical analyses

Conditional logistic regression will be used to estimate odds ratios (ORs) and corresponding 95% confidence intervals (CIs) of the association of hospitalization for AP, comparing incretin-based drugs to current use of oral anti-diabetic drug combinations. This is considered the primary analysis. Secondary analyses will include sub-classifying current users of incretin-based drugs by type (i.e., DPP-4 inhibitor vs GLP-1 analog) and duration of current use (≤ 365 days, 366-729 days, and ≥730 days). The potential presence of effect modification by history of acute pancreatitis will also be examined. In addition, seven sensitivity analyses will be conducted; all defined a priori, to assess the robustness of the results. Finally, all site-specific estimates will be meta-analyzed using random-effects models with inverse variance weighting, with fixed-effects analyses conducted as sensitivity analyses. The amount of between-site heterogeneity will be estimated using the I square statistic.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a first-ever prescription for a non-insulin anti-diabetic drug, including biguanides, sulfonylureas, thiazolidinediones, DPP-4 inhibitors, GLP-1 analogs, alpha-glucosidase inhibitors, meglitinides or combinations of these drugs from the earliest availability of data at each site to the last date of availability of data.
* Patients with at least 1 year of history in the database.
* Patients at least 18 years of age.

Exclusion Criteria:

* Patients who died or left the cohort before the year the first incretin-based drug entered the market.
* Patients who never added-on or switched to a new anti-diabetic drug after incretin-based drugs entered the market up until June 30, 2014.
* Patients with a previous diagnosis of pancreatic cancer, those who underwent pancreatectomy, those with diagnoses of congenital defects of the pancreas, cystic fibrosis, lupus, or previous bariatric surgery, at any time prior to study cohort entry.
* Patients diagnosed with HIV or initiating HAART therapy before and at study cohort entry.
* Patients hospitalized for acute pancreatitis in the 30 days before study cohort entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In each jurisdiction, the investigators will assemble a base cohort including all patients with a first-ever prescription for a non-insulin anti-diabetic drug. Base cohort entry is defined as the date of prescription or dispensation of the first-ever non-insulin anti-diabetic drug. From this base cohort, a study cohort will be formed including all patients who initiated a new anti-diabetic drug class during the year in which incretin-based drugs entered the market in each jurisdiction or any time thereafter. Study cohort entry is defined by the prescription date of the newly-prescribed drug class.
Sampling Method: Probability Sample
Enrollment: 1417914 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Hospitalization for acute pancreatitis | Patients were followed from the date of study cohort entry until hospitalization for incident acute pancreatitis, censoring, or for up to 87 months.
  Incident hospitalization for acute pancreatitis recorded in either physician or hospital databases with the following ICD codes:
  ICD-9: 577.0 ICD-10: K85.0, K85.1, K85.2, K85.3, K85.8, and K85.9 in the primary [or most responsible] or secondary position, including post-admission diagnoses)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Ernst, MD, MSc, Principal Investigator — Lady Davis Institute for Medical Research, Jewish General Hospital - McGill University
Locations (1):
- Lady Davis Institute for Medical Research, Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Result] Azoulay L, Filion KB, Platt RW, Dahl M, Dormuth CR, Clemens KK, Durand M, Hu N, Juurlink DN, Paterson JM, Targownik LE, Turin TC, Ernst P; and the Canadian Network for Observational Drug Effect Studies (CNODES) Investigators; Suissa S, Dormuth CR, Hemmelgarn BR, Teare GF, Caetano P, Chateau D, Henry DA, Paterson JM, LeLorier J, Levy AR, Ernst P, Platt RW, Sketris IS. Association Between Incretin-Based Drugs and the Risk of Acute Pancreatitis. JAMA Intern Med. 2016 Oct 1;176(10):1464-1473. doi: 10.1001/jamainternmed.2016.1522. PMID 27479930
- See also: This organization's website describing general functions, other CNODES projects, and investigator profiles. — http://www.cnodes.ca